CLINICAL TRIAL: NCT03936881
Title: Attitude of the Dentist to the Detection of Calcification of the Carotid Region on an Orthopantomogram
Brief Title: Carotid Region Calcifications and Orthopantomogram
Acronym: ADCACO
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_30024_ADCACO
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study.

DETAILED DESCRIPTION:
The orthopantomogram or dental panoramic is a routine screening examination in dental practice. It is defined as a two-dimensional, inexpensive examination that provides an overview of bone and dental structures, temporomandibular joints, nasal cavities and maxillary sinuses. While the dentist's attention is focused primarily on dento-maxillary structures, careful examination of the dentist may reveal radiopaque images in the submandibular region, which Friedlander calls the Carotid Artery Territory and defines as the projection region of the common carotid artery, the carotid bifurcation and the internal carotid artery. Calcifications observed at this level can be of two types: anatomical and pathological. Among the so-called pathological calcifications are the calcifications of the carotid artery which are described in the literature as irregular, appearing as vertical, heterogeneous, uni- or bilateral lines and located at the angle of the mandible opposite C3-C4. A table was proposed by Pornprasertsuk-Damrongsri in 2006 allowing the differential diagnosis of these calcifications of the carotid artery with other types of calcifications based on an exhaustive a priori analysis of the literature.

The radiopacities identified as carotid calcifications are in fact calcifications that appear on a prior thickening of the vascular wall of a carotid artery corresponding to an atheroma plaque. This atheroma plaque can generate occlusions (such as embolism or stenosis).

In addition, some studies have shown a correlation between the detection of carotid artery calcifications from the orthopantomogram and the presence of Doppler stenosis. Currently the Doppler is the gold standard test for diagnosing carotid stenosis.

Romano-sousa in its 2009 study shows a strong correlation between the detection of carotid calcifications on the orthopantomogram and Doppler images: calcifications are observed on both the orthopantomogram and Doppler in 59.4% of cases. Almog (2002) finds 50% stenosis (>50%) in analyzed sides with calcifications; compared to 21% in sides where there is no calcification.

In 1998, Friedlander concluded that dentists could have a role in preventing cardiovascular events by screening carotid artery calcifications on the orthopantomogram, and included this analysis of the orthopantomogram in a public health approach that would reduce mortality and morbidity from ischemic stroke, as well as the costs associated with lost productivity, hospitalization and rehabilitation. Indeed, stroke is the third leading cause of death in developed countries and a major cause of serious morbidity.

It therefore seems interesting to be able to detect asymptomatic carotid stenosis in order to implement an appropriate diagnostic and therapeutic strategy. On the other hand, the accidental discovery of carotid artery calcifications on an orthopantomogram indicates a general arterial abnormality. It may therefore be interesting to detect possible calcifications of the carotid artery in middle-aged patients with no cardiovascular history or risk factors for cardiovascular events.

On the other hand, some authors mention a link between the presence of calcifications of the carotid artery and the existence of periodontal disease. Indeed, both are linked to an inflammatory phenomenon. The investigators will therefore try to see if this relationship exists in the investigator's population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years of age or older) attending the dental care centre at the Rennes University Hospital;
* Who had an orthopantomogram radiological examination at the Rennes Dental Care Centre between 1 September 2018 and 31 December 2018;
* Having agreed to the use of its data for teaching or publication purposes.

Exclusion Criteria:

* Orthopantomogram not usable, not allowing to visualize the sub-mandibular region (due to poor patient positioning);
* Persons of full age who are subject to legal protection (protection of justice, guardianship, guardianship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who presented themselves at the Dental Care Centre of the Rennes University Hospital between 1 September 2018 and 31 December 2018
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Presence or absence of calcifications of the carotid area | During the realization of the orthopantomogram (between 1 September 2018 and 31 December 2018)
  Calcifications of the carotid as recorded on the orthopantomogram of the patient

SECONDARY OUTCOMES:
Presence or absence of a cardiovascular pathology | During the consultation at the Dental Care Centre (between 1 September 2018 and 31 December 2018)
  Cardiovascular pathology as recorded on the medical record of the patient.
Presence or absence of moderate to severe alveolysis | During the consultation at the Dental Care Centre (between 1 September 2018 and 31 December 2018)
  Periodontal disease as recorded during the consultation at the dental centre

CONTACTS AND LOCATIONS:
Overall Officials: Guy CATHELINEAU, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France